CLINICAL TRIAL: NCT04101253
Title: SCREENING FOR THE IMPLANTATION OF A SUBCUTANEOUS IMPLANTABLE AUTOMATIC DEFIBRILLATOR: OPTIMIZATION OF THE PROCEDURE BY REPOSITIONING THE ELECTRODES AND RESEARCH OF THE PREDICTIVE FACTORS OF FAILURE
Brief Title: SCREENING FOR THE IMPLANTATION OF A SUBCUTANEOUS IMPLANTABLE AUTOMATIC DEFIBRILLATOR
Acronym: SIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de PAU (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHPAU2019/02
Record Dates: First submitted 2019-09-19; First posted 2019-09-24 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Sudden Cardiac Death; Implantable Defibrillator
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Every ICD patient will undergo the standard screening process. Initial screening will be performed as usually performed by physician or Boston Scientific technical support. In case of one or more vector satisfying screening criteria, patient will be assigned in "screening success" group. In case of failure, a pre-determined electrode positioning protocol will be done with variation of para-sternal and axillary electrodes. Positioning variations will be left to the discretion of the operator cardiologist.
  Interventions: Procedure: new screening procedure with small variations in electrode positioning

INTERVENTIONS:
Procedure: new screening procedure with small variations in electrode positioning — Every ICD patient will undergo the standard screening process. Initial screening will be performed as usually performed by physician or Boston Scientific technical support. In case of one or more vector satisfying screening criteria, patient will be assigned in "screening success" group. In case of failure, a pre-determined electrode positioning protocol will be done with variation of para-sternal and axillary electrodes. Positioning variations will be left to the discretion of the operator cardiologist.

SUMMARY:
S-ICD (subcutaneous implantable cardioverter-defibrillator) screening failure occurs in about 10% of cases. Predictors of screening failure are not yet well determined. Moreover, slight variations in electrode positioning may change vector configuration and therefore improve screening success rates

DETAILED DESCRIPTION:
S-ICD (subcutaneous implantable cardioverter-defibrillator) has become the last years widespread in various pathological conditions and implantation rates are increasing each year worldwide. Previous to implantation it is mandatory to realize a screening in order to assess specific electrocardiographic vectors used to analyze cardiac rhythm. In routine practice, approximatively 10% of patients are recused for S-ICD device implantation due to failed screening 1-3. Causes are mainly abnormalities of R wave (low or high amplitude) and low R/T wave ratio. Determinants for screening failure have not yet been clearly studied. Moreover, it is a common finding in S-ICD implantation to find variations between pre-implant electrograms and electrograms recorded by the device. Variations of R wave amplitude and R/T ration are also observed with small variations of electrode positioning prior to implantation. It has been also shown that despite initial screening failure, S-ICD could be securely performed in some cases 4,5. Patients included in the study will undergo usual screening protocol. In case of failure a 2nd screening will be realize with slight electrode positioning variations compatible with S-ICD and lead placement. In case of success modality of implantation will be decided by physician.

In case of S-ICD implantation screening data will be compared to post implantation device electrograms. A 2 month follow-up will be performed with comparison of a new screening procedure with electrodes at the level of sub-cutaneous electrodes.

ELIGIBILITY:
Inclusion Criteria:

* The population will be composed of all patients referred for ICD method, aged over 18 years

Exclusion Criteria:

* Age < 18 years old
* Patients who cannot freely give their consent, or patients who refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
screening success rates | one day
  Comparison of success rates between the standard screening procedure (without repositioning the electrodes) and the proposed new procedure (small variations in electrode positioning)

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - CHRU de BREST, Brest
  - CHU de Caen, Caen
  - CHRU de Lille, Lille
  - Hopital Saint Philivert, Lille
  - CHU de Limoges, Limoges
  - Hopitl Cardiologique Louis Pradel, Lyon
  - CHU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - AP-HP Hôpital européen Georges-Pompidou, Paris
  - APHP - Pitié Salpêtrière, Paris
  - CH de Pau, Pau
  - CHU de Rennes, Rennes
  - CHRU de Strasbourg, Strasbourg
  - CHU deToulouse, Toulouse
  - Clinique Pasteur, Toulouse
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Guillebon M, Garcia R, Debeugny S, Bader H, Probst V, Bidegain N, Narayanan K, Mansourati J, Menet A, Ollitrault P, Marquie C, Guy-Moyat B, Mondoly P, Chevalier P, Badenco N, Behar N, Jesel-Morel L, Pierre B, Lellouche N, Deharo JC, Jacon P, Anselme F, Boveda S, Marijon E; SIS Study Investigators. Personalized screening before subcutaneous cardioverter-defibrillator implantation: Usefulness and outcomes in clinical practice-the S-ICD screening SIS prospective study. Heart Rhythm. 2024 Dec;21(12):2530-2535. doi: 10.1016/j.hrthm.2024.05.043. Epub 2024 May 27. PMID 38810921